CLINICAL TRIAL: NCT07212959
Title: CXCR4-PET/CT for the Detection of Inflammatory Activity in Systemic Sclerosis
Brief Title: As Part of a Pilot Study, Visualization of Inflammatory Activity in Systemic Sclerosis Using CXCR4 PET/CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 296/21-me
Record Dates: First submitted 2025-10-02; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Systemic Sclerosis (SSc)
Keywords: SSc; CXCR4; PET/CT
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CXCR4-PET/CT for detection von inflammatory changes in systemic sclerosis (Experimental)
  Interventions: Other: CXCR4-PET/CT

INTERVENTIONS:
Other: CXCR4-PET/CT — CXCR4-PET/CT for the detection of inflammatory activity in patient with active systemic sclerosis

SUMMARY:
Systemic sclerosis (SSc) is a heterogeneous clinical picture consisting of inflammatory, vasculopathic, and fibrotic changes.

Initially, inflammatory changes usually occur, which result in fibrosis over time.

This affects various organ systems such as the lungs, skin, heart, and gastrointestinal tract. Early detection of inflammatory activity is therefore important in order to prevent consequential damage, in particular irreversible fibrosis. Since the inflammatory foci can spread throughout the entire body, there is a need to be able to detect inflammatory activity over a large area. The 68Ga-Pentiafor-based imaging of the CXCR4 chemokine receptor, which is expressed on immune system cells such as lymphocytes and macrophages, among others, offers a useful approach here, as it allows specific inflammatory cells that migrate to inflammatory lesions via the corresponding ligand (CXCL12) and are involved in the pathogenesis of SSc. To date, only chest CT has been used to diagnose and monitor the progression of pulmonary fibrosis in SSc. This non-functional imaging makes it virtually impossible to draw conclusions about inflammatory activity.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SSc based on the 2013 ACR/EULAR criteria
* Duration of disease less than 5 years (onset of the first non-Raynaud's symptom within the last 5 years)
* Evidence of ILD on computed tomography
* Patient's ability to understand the information provided
* Patient of legal age

Exclusion Criteria:

* Following autologous stem cell transplantation
* Presence of pulmonary hypertension
* Contraindications for performing a PET/CT scan - Pregnancy
* Breastfeeding
* Allergies to 68Ga-Pentixafor
* Patient's inability to understand and give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Maximum Traceracktivity in CXCR4-PET/CT | 2 year
  Measurement of the maximum measurable CXCR4 tracer activity in CXCR4 PET/CT in fibrotic pulmonal changes

CONTACTS AND LOCATIONS:
Overall Officials: MIcheal Armin Gernert, Privatdozent, Study Director — Wuerzburg University Hospital
Locations (1):
- University Hospital Würzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT07212959/Prot_000.pdf